CLINICAL TRIAL: NCT03233048
Title: Safety and Efficacy of Endoscopically Placed Intragastric Balloon in Obese Adolescents With Comorbidities - A Pilot Study
Brief Title: Intragastric Balloon in Obese Adolescents With Comorbidities
Acronym: IGB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imad Absah (Other)
Responsible Party: Sponsor-Investigator, Imad Absah, Assistant Professor of Pediatrics, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-009191
Record Dates: First submitted 2017-07-26; First posted 2017-07-28 (Actual); Results first posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ORBERA™ Intragastric Balloon (Experimental): Participants will have the ORBERA™ Intragastric Balloon inserted for 6 months. In addition, participants will have ongoing visits with a physician, dietitian, and psychologist before the balloon is inserted, while its in place, and for 6 months after the balloon is removed, for a total of approximately 1 year.
  Interventions: Device: ORBERA™ Intragastric Balloon

INTERVENTIONS:
Device: ORBERA™ Intragastric Balloon — The balloon will be inserted into the stomach and inflated, and will remain in place for 6 months, after which the device will be removed.

SUMMARY:
The reason we are doing this research is to get information about the ORBERA™ Intragastric Balloon to learn if it is safe and if it works. We want to learn if older teenagers who are overweight will lose weight and if their other medical problems will get better. ORBERA™ is a special balloon approved by the FDA for overweight adults, and we would like to try using it for overweight teenagers.

DETAILED DESCRIPTION:
After obtaining consent and determining that participants meet the inclusion and exclusion criteria, participants will have baseline tests and initial visits with a physician, dietitian, and psychologist. Next, the ORBERA™ Intragastric Balloon (IGB) will be inserted into the stomach and then removed after 6 months. Participants will continue to be followed for 6 months after the balloon is removed. Throughout the year, participants will have additional tests along with ongoing visits with a physician, dietitian, and psychologist.

ELIGIBILITY:
Inclusion Criteria:

BMI>35 kilogram per square meter (kg/m2) with one of the following severe comorbidities, both for at least 2 years:

1. Type 2 diabetes mellitus
2. Moderate-to-severe sleep apnea
3. Pseudotumor cerebri
4. Nonalcoholic Steatohepatitis (NASH) based on fatty infiltration of the liver with transaminitis that cannot be explained by other liver disease

Or,

BMI>40 kilogram per square meter (kg/m2) with two or more of the following mild comorbidities, all for at least 2 years:

1. Hypertension
2. Dyslipidemia
3. Mild obstructive sleep apnea
4. Chronic venous insufficiency
5. Panniculitis
6. Urinary incontinence
7. Nonalcoholic Steatohepatitis (NASH)
8. Gastroesophageal reflux disease (GERD)
9. Arthropathies related to weight

In addition, all of the following inclusion criteria must be met. The subject must have:

1. attained approximately 95% of adult stature, as demonstrated by Tanner Stage IV or more and growth charts demonstrating the taper/plateau of height as a marker for achieving 95% of the subject's adult stature. Height will be measured by trained staff to the nearest 0.1 cm using a stadiometer attached to a wall and documented in the subject's electronic medical record (EMR). In the absence of previous growth charts, skeletal maturity will be documented by a bone age of at least 13 years in girls and 15 years in boys; and
2. failed to attain a healthy weight with at least one experience with medically supervised lifestyle changes, including physical activity and dietary interventions, which will be clearly documented in the subject's medical record, and
3. demonstrated commitment to psychological evaluation perioperatively, in which the pediatric psychologist with expertise in childhood obesity must confirm that the subject has the maturity and stable psychosocial environment necessary for this research study and has validated the Center for Epidemiology Study Depression (CES-D) scale and Spence Children's Anxiety Scale (SCAS) surveys completed by the subject, and
4. agreed to avoid pregnancy for 1 year after intragastric balloon (IGB) placement through abstinence or approved contraception (female subjects only), and
5. agreed to adhere to nutritional guidelines after intragastric balloon (IGB) placement, as provided by weight management clinic dietitian, and
6. decisional capacity and desire to provide informed assent in conjunction with parent/guardian consent, and willingness to comply with all study requirements, and
7. hypertension stage I: systolic blood pressure and/or diastolic blood pressure ≥ 95th percentile, OR high normal blood pressure between the 90th and 95th percentile.

Exclusion Criteria:

Subjects will be excluded if:

1. they are pregnant or breastfeeding, or
2. there is any other disease, physical examination finding, or clinical laboratory result that provides a reasonable suspicion of a disease or condition that contraindicates the use of the investigational device or that may affect the interpretation of the results or render the subject at high risk for treatment complications, or
3. there is alcohol, tobacco, or substance use by the subject, or
4. in the opinion of the principal investigator (PI) and/or co-investigators, subject or parent/guardian may be non-compliant with study schedules or procedures, or
5. there are any endoscopic contraindications, including large hiatal hernia (≥ 2 cm), esophagitis of any degree, erosive gastritis, or ulceration of the stomach or duodenum, or
6. Helicobacter pylori (H. pylori) is detected via a fecal antigen study prior to initial endoscopic assessment (sensitivity > 96.8%); once treated, a repeat fecal antigen must be performed to document eradication prior to the first endoscopic approach for balloon placement, or
7. they have hypertension stage II > 99th percentile, unless they had a complete workup to exclude secondary etiologies other than being overweight, or
8. Gastroesophageal reflux disease (GERD) subjects are on more than one medication or have a history of erosive esophagitis due to gastroesophageal reflux disease (GERD), or
9. they have dyslipidemia, if part of hereditary metabolic syndrome or genetic disorder, or
10. they have any gastrointestinal disease that can result in stomach ulcerations, such as Crohn's disease, celiac disease, eosinophilic esophagitis, acute or chronic pancreatitis or gastrinoma, or
11. they have any endocrine disorders that affect metabolic status of the subjects, such as hypo/hyperthyroidism, type 1 diabetes, Cushing's disease, or adrenal insufficiency, as documented in the electronic medical record (EMR) through an evaluation by the pediatric endocrinologist who will order additional testing if needed, or
12. they have prior gastrointestinal surgery with sequelae, i.e. obstruction, and/or adhesive peritonitis or known abdominal adhesions and/or history of abdominal and/or pelvic surgery which may cause adhesions (except one of the following: caesarean section, diagnostic laparoscopy, laparoscopic appendectomy, laparoscopic cholecystectomy performed 12 or more months prior to balloon implantation), or
13. they have prior open or laparoscopic bariatric surgery, or
14. they have prior surgery of any kind on the esophagus, stomach or any type of hiatal hernia surgery, or
15. they have any inflammatory disease of the gastrointestinal tract including esophagitis, Barrett's esophagus, cancer or specific inflammation such as Crohn's disease, or
16. they have potential upper gastrointestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasis, or other congenital anomalies of the gastrointestinal tract such as atresias or stenoses, or,
17. they have a gastric mass, or
18. they have acid reflux symptoms to any degree that require more than one medication for symptom control, or
19. they have a structural abnormality in the esophagus or pharynx such as a stricture or diverticulum that could impede passage of the balloon alongside the endoscope, or
20. they have achalasia or any other severe esophageal motility disorder that may pose a safety risk during the removal of the device, or
21. they have severe coagulopathy, or
22. they have poorly controlled diabetes, defined as having a Hemoglobin A1c (HgA1c) > 10, or
23. they have serious health conditions unrelated to their weight that would increase the risk of endoscopy, or
24. they have chronic abdominal pain, or
25. they have motility disorders of the gastrointestinal (GI) tract such as gross esophageal motility disorders, gastroparesis, or intractable constipation, or
26. they have hepatic insufficiency or cirrhosis, or
27. they have serious or uncontrolled psychiatric illness or disorder that could compromise their understanding of, or compliance with, follow-up visits and removal of the device, or
28. they are receiving daily prescribed treatment with aspirin, anti-inflammatory agents, anticoagulants or other gastric irritants, or
29. they are taking medications on specified hourly intervals that may be affected by changes to gastric emptying, such as anti-seizure or anti-arrhythmic medications, or
30. they are taking corticosteroids, immunosuppressants, or narcotics, or
31. they are unable or unwilling to take prescribed proton pump inhibitor medication, or
32. they are known to have, or suspected to have, an allergic reaction to materials contained in the system, or
33. they have ever developed a serotonin syndrome and are currently taking any drug known to affect the levels of serotonin in the body (e.g. selective serotonin reuptake inhibitors, serotonin-norepinephrine reuptake inhibitors, monoamine oxidase inhibitors), or
34. they have a medically identifiable cause of obesity (specific diagnosed genetic or hormonal case for obesity such as hypothyroidism or Prader Willi syndrome), or
35. they have known history of endocrine disorders affecting weight, or
36. they use any medications, except for Metformin, known to affect body weight and carbohydrate or lipid metabolism, or
37. they used an intragastric device prior to this study, or
38. they participated in any clinical study which could affect weight loss within the past 6 months, or
39. they have symptomatic congestive heart failure or cardiac arrhythmia, or
40. they have a diagnosis of an autoimmune connective tissue disorder (e.g. lupus, erythematous, scleroderma), or immunocompromised, or
41. they are on insulin for type 2 diabetes and not proficient in self-monitoring capillary blood glucose testing.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Absah, M.D., Principal Investigator — Study Principal Investigator
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ORBERA™ Intragastric Balloon
Started | 5
Completed | 4
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Achieving Greater Than or Equal to 10% Total Body Weight Loss
Description: Weight loss will be measured by change in weight divided by baseline weight.
Time Frame: up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
Participants | 2

2. Secondary Outcome: Change in Alanine Aminotransferase (ALT)
Description: Change will be measured as a percentage by taking change in ALT divided by baseline ALT.
Time Frame: Baseline, end of study (approximately 1 year)
Measure: Mean (Standard Deviation); unit: percentage of change in ALT level
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
percentage of change in ALT level | 25.7 (36)

3. Secondary Outcome: Change in Aspartate Aminotransferase (AST)
Description: Change will be measured as a percentage by taking change in AST divided by baseline AST.
Time Frame: Baseline, end of study (approximately 1 year)
Measure: Mean (Standard Deviation); unit: percentage of change in AST level
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
percentage of change in AST level | 11.5 (12)

4. Secondary Outcome: Change in Fasting Insulin
Description: Change will be measured as a percentage by taking change in fasting insulin divided by baseline fasting insulin.
Time Frame: Baseline, end of study (approximately 1 year)
Measure: Mean (Standard Deviation); unit: percentage of change in insulin level
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
percentage of change in insulin level | 33 (57.5)

5. Secondary Outcome: Change in Hemoglobin A1c (HgA1c)
Description: Change will be measured as a percentage by taking change in HgA1c divided by baseline HgA1c.
Time Frame: Baseline, end of study (approximately 1 year)
Measure: Mean (Standard Deviation); unit: percentage of change in HgA1c level
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
percentage of change in HgA1c level | 0.5 (0.3)

6. Secondary Outcome: Change in High-density Lipoprotein (HDL)
Description: Change will be measured as a percentage by taking change in HDL divided by baseline HDL.
Time Frame: Baseline, end of study (approximately 1 year)
Measure: Mean (Standard Deviation); unit: percentage of change in HDL level
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
percentage of change in HDL level | 23.4 (31)

7. Secondary Outcome: Change in Low-density Lipoprotein (LDL)
Description: Change will be measured as a percentage by taking change in LDL divided by baseline LDL.
Time Frame: Baseline, end of study (approximately 1 year)
Measure: Mean (Standard Deviation); unit: percentage of change in LDL level
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
percentage of change in LDL level | 9 (19)

8. Secondary Outcome: Change in Triglycerides
Description: Change will be measured as a percentage by taking change in triglycerides divided by baseline triglycerides.
Time Frame: Baseline, end of study (approximately 1 year)
Measure: Mean (Standard Deviation); unit: percentage of change in triglycerides
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
percentage of change in triglycerides | 28 (22)

9. Secondary Outcome: Number of Participants With One or More Serious Adverse Events
Description: Number of participants to experience one or more serious adverse events as defined as Grade 3 or higher according to Common Terminology Criteria for Adverse Events (CTCAE) scale.
Time Frame: Intragastric balloon (IGB) removal (approximately 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
Participants | 0

10. Secondary Outcome: Number of Subjects Who Had the Balloon Removed Early
Description: Early will be defined as balloon removal prior to the 6 month window time point as defined in the protocol.
Time Frame: Intragastric balloon (IGB) removal (approximately 6 months)
Population: At the request of the subject Intragastric balloon (IGB) was removed at 3 months and the subject was withdrawn from the study (withdrawal by subject).
Measure: Count of Participants; unit: Participants
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 5
Participants | 1

11. Secondary Outcome: Number of Subjects Whose Balloon Deflated Early
Description: Early will be defined as balloon deflation prior to the 6 month window time point as defined in the protocol.
Time Frame: Intragastric balloon (IGB) removal (approximately 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | ORBERA™ Intragastric Balloon
Number analyzed (Participants) | 4
Participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 12 months on all participants
Arm/Group | ORBERA™ Intragastric Balloon
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORBERA™ Intragastric Balloon (N=5)
Nausea (Gastrointestinal disorders) | 3 (3)
Abdominal pain/discomfort (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT03233048/Prot_SAP_000.pdf